CLINICAL TRIAL: NCT06923020
Title: Exploring the Correlation Between Nutritional Status and Efficacy of First-Line Immune Checkpoint Inhibitors in Metastatic Esophagogastric Cancer: A Prospective Cohort Study.(Nutrition EGC)
Brief Title: Association of Nutritional Status With Immune Checkpoint Inhibitor Efficacy in Metastatic Metastatic Esophagogastric Cancer.
Status: Enrolling by invitation | Type: Observational
Sponsor: Yongxu Jia (Other)
Responsible Party: Sponsor-Investigator, Yongxu Jia, The First Affiliated Hospital of Zhengzhou University, The First Affiliated Hospital of Zhengzhou University
Organization: The First Affiliated Hospital of Zhengzhou University (Other)
Other Study IDs: Nutrition EGC-2024-KY-002
Record Dates: First submitted 2025-04-09; First posted 2025-04-11 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2025-04

CONDITIONS: Gastric Neoplasm; Esophageal Adenosquamous Carcinoma
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Cohort A: advanced GC patients receiving first-line ICIs
  Interventions: Other: Exposure: Nutritional Status
- Cohort B: advanced ESCC patients receiving first-line ICIs
  Interventions: Other: Exposure: Nutritional Status

INTERVENTIONS:
Other: Exposure: Nutritional Status — The assessment of nutritional risk screening (NRS) and nutritional assessments were conducted using NRS 2002 and Patient-Generated Subjective Global Assessment (PG-SGA).
  Groups: Cohort A
Other: Exposure: Nutritional Status — The assessment of nutritional risk screening (NRS) and nutritional assessments were conducted using NRS 2002 and Patient-Generated Subjective Global Assessment (PG-SGA).
  Groups: Cohort B

SUMMARY:
In patients with advanced gastrointestinal cancers, malnutrition can lead to increased incidence of adverse events during the peri-chemoradiotherapy period, reduced treatment tolerance, lower completion rates of therapy, compromised efficacy and quality of life, and ultimately shortened survival. Currently, immunotherapy represented by PD-1 inhibitors has become a cornerstone in the treatment of advanced gastrointestinal cancers. Nutritional status plays a critical role in malignancies, with the Prognostic Nutritional Index (PNI) and Controlling Nutritional Status (CONUT) score being particularly important for assessing nutritional conditions in cancer patients. Gastrointestinal cancers, as a group of heterogeneous tumors with distinct morphological and molecular genetic features, are closely linked to nutritional status. Peripheral blood cell profiles reflect the inflammatory impact of malignancies and immune responses in patients, which are crucial for determining treatment responses and clinical outcomes to enable early stratification, intervention, and monitoring. Therefore, this study aims to explore the clinical significance of nutrition-related prognostic indicators in immunotherapy by evaluating nutritional status and comparing treatment efficacy of first-line immune checkpoint inhibitors among advanced gastric cancer and esophageal cancer patients (including unresectable locally advanced, recurrent, or metastatic gastrointestinal cancers such as gastric/gastroesophageal junction adenocarcinoma and esophageal carcinoma) with different nutritional profiles.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed esophageal squamous carcinoma and gastric adenocarcinoma, metastatic disease.
* Measurable disease according to the RECIST criteria(diameter of the lesion should be more than 10mm by spiral CT or MRI, more than 20mm by common CT, the date of image should be less than 15 days before enrollment)
* Karnofsky performance status ≥80
* Life expectancy of ≥ 3 month
* WBC > 3,000/mm3, absolute neutrophil count ≥1500/mm3, platelet > 100,000/mm3, Hb > 9g/dl(within 14 days before enrollment),ALT and AST < 2.5 times ULN (≤5 times ULN in patients with liver metastases),Bilirubin level < 1.0 times ULN,Serum AKP < 2.5 times ULN,Serum creatinine < 1.5 times ULN
* No sever complication, such as active gastrointestinal bleeding, perforation, jaundice, obstruction, non-cancerous fever > 38℃；
* Normal ECG and heart function
* Fertile patients must use effective contraception
* Good compliance

Exclusion Criteria:

* Previous treatment of palliative chemotherapy
* Only with Brain or bone metastasis
* No measurable lesions, eg. pleural fluid and ascites
* Suffer from severe heart disease or disease with other important organs
* Chronic diarrhea or renal dysfunction
* Pregnancy or lactation period
* Other previous malignancy within 5 year, except non-melanoma skin cancer Chronic diarrhea
* Mentally abnormal or disable cognition,including CNS metastasis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: metastatic ESCC and GC patients receiving the first-line therapy ICIs
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-10-31 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2027-10-31 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) | 5 years
  Overall survival (OS) is defined as the duration from the beginning of first-line immunotherapy until death due to any cause. Subjects who are still alive at the end of the study observation period will be censored at the time of last known vital status.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | 3 years
  Time from the beginning of first-line immunotherapy to the first progression (PD) in patients with EGC.

CONTACTS AND LOCATIONS:
Locations (1):
- Yongxu Jia, Zhengzhou, Henan, China